CLINICAL TRIAL: NCT06658171
Title: Effects of Relaxation Training and Stimulus Control in Chronic Insomnia Patients With Hyperarousal and Maladaptive Sleep Patterns
Brief Title: Effects of Relaxation Training and Stimulus Control in Chronic Insomnia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT-SC-insomnia
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Chronic Insomnia
Keywords: chronic insomnia; sleep restriction; stimulus control; sleep hygiene education
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Relaxation training and stimulus control (Experimental)
  Interventions: Behavioral: Relaxation training and stimulus control
- Sleep hygiene education (Active Comparator)
  Interventions: Behavioral: Sleep hygiene education

INTERVENTIONS:
Behavioral: Relaxation training and stimulus control — Relaxation training: Progressive muscle relaxation; Breathing relaxation; Imagery training; Mindfulness relaxation.
  Stimulus control: a) Reduce wakeful time in bed and rebuild a positive association between sleepiness and bed; b) Use the bed solely for sleeping and sexual activities; c) Only go to bed when feeling sleepy at night or at the designated sleep time; d) If unable to fall asleep within about 20 minutes of being in bed, leave the bedroom and engage in relaxation activities until feeling sleepy, then return to bed for sleep; if still unable to fall asleep within about 20 minutes, repeat the process; e) Wake up at the same time every morning, including weekends.
  Arms: Relaxation training and stimulus control
Behavioral: Sleep hygiene education — 1. Sleep until feeling refreshed the next day.
  2. Maintain regular exercise and eating habits, avoiding going to bed on an empty stomach.
  3. Ensure a comfortable bedroom environment with suitable nighttime temperature, free from light and noise disturbances.
  4. Avoid excessive consumption of beverages, alcohol, and smoking at night, and reduce caffeine intake.
  5. Avoid bringing problems to bed and refrain from attempting to sleep.
  6. Place the alarm clock under the bed or move it away from sight.
  7. Avoid daytime napping.
  Arms: Sleep hygiene education

SUMMARY:
The study aims to validate the effect of relaxation training and stimulus control on reducing hyperarousal states and improving maladaptive sleep behaviors.

DETAILED DESCRIPTION:
Relaxation training typically includes techniques such as breathing exercises, muscle relaxation, and mindfulness meditation to help patients reduce levels of physical and psychological tension, promote relaxation, and create favorable conditions for sleep onset. Stimulus control aims to break the negative association between the bed and insomnia, and rebuild a positive association between the bed and sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for insomnia disorder according to DSM-5.
2. Pittsburgh Sleep Quality Index (PSQI) total score > 5.
3. Age ≥ 18 years, with at least a middle school education level.
4. Anxiety symptoms meeting HAMA ≥ 14.
5. "Self-developed 8-item questionnaire on maladaptive sleep behaviors" used to assess "maladaptive sleep behaviors."
6. Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Individuals with severe physical illnesses or severe mental disorders, at risk of suicide.
2. Clinically diagnosed or suspected sleep-related breathing disorders, restless leg syndrome, and sleep-wake rhythm disorders, as well as shift workers.
3. Pregnant or lactating women.
4. Currently undergoing any psychological therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The change of Pittsburgh Sleep Quality Index (PSQI) total scores from baseline to 6 weeks. | Baseline, 6 weeks
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.

SECONDARY OUTCOMES:
The change of PSQI total scores from baseline to 3 months, 6 months, and 12 months. | Baseline, 3 months, 6 months, and 12 months
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.
The change of Insomnia severity index (ISI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The ISI reporting insomnia symptoms severity consists of 7-items on a 5-point Likert scale, and the total score ranges from 0 to 28 with higher scores indicating more severe insomnia.
The change of sleep efficiency from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  Sleep efficiency is assessed with the Carney (2012) consensus sleep diary. This is measured in percentage (higher scores indicating better sleep efficiency).
The change of Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The DBAS assessing sleep related cognitions in 16 items rated on a 10-point Likert scale, and the total score ranges from 0 to 160 with higher scores indicating more intensive dysfunctional beliefs.
The change of Snaith-Hamilton Pleasure Scale (SHAPS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The SHAPS assessing anhedonia consists of 14 items, and the total score ranges from 14 to 56 with higher scores indicating more serious the anhedonia.
The change of Short Form 36 (SF-36) total scores from baseline to 6 weeks, 3 months, 6 months, 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months.
  The SF-36 quantifying the quality of life in relation to health status consists of 36-items with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The total score ranges from 0-100 (the worst possible to the most possible).
The change of Patient Health Questionnaire-4 (PHQ-4) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-4 comprises a 2-item depression scale and a 2-item anxiety scale. Each instrument can reach values from 0-6. Higher Scores are indicating higher distress.
The change of Beck Depression Inventory (BDI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BDI assessing the existence and severity of symptoms of depression consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe depressive symptoms.
The change of Beck Anxiety Inventory (BAI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BAI assessing the existence and severity of symptoms of anxiety consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe anxiety.
The change of Patient Health Questionnaire-15 (PHQ-15) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-15 measuring somatic distress consists of 15 items, and the total score ranges from 0 to 30 with higher scores indicating more severe somatic distress.
The change of 5-item Perceived Deficits Questionnaire-Depression (PDQ-D-5) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PDQ-D-5 assessing perceived cognitive deficits from the patient's perspective consists of 5 items, and the total score ranges from 0 to 20 with higher scores indicating greater perceived deficit.
The change of Life Events Scale (LES) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The LES assessing the perceived stress and number of stressful life events experienced consists of 48 items which are classified into three dimensions: family life events (28 items), work and study events (13 items), and social events (7 items) with higher scores in LES perceived greater stressfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China